CLINICAL TRIAL: NCT05744947
Title: Modalities And Safety Of Cardiac Rehabilitation In A Population Managed For Spontaneous Hematoma Or Coronary Disruption (DISCO): Data From The DISCO Study
Brief Title: Modalities And Safety Of Cardiac Rehabilitation In A Population Managed For Spontaneous Hematoma Or Coronary Disruption
Acronym: READAPT-DISCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/52
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Rehabilitation Program Following the Management of ACS in Patients Presenting With SCAD
Keywords: Cardiac rehabilitation; Spontaneous Coronary Artery Dissection
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recruited patient .: Patient previsouly recruited in the DISCO Registry (Study of the Prevalence Fibromuscular Dysplasia in Patient With Haematoma or Spontaneous Coronary Artery Dissection. (DISCO trial - NCT02799186)) with cardiac rehabilitation following the management of acute coronary syndrome
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Specific "Readapt -DISCO" complementary questionnaire rehabilitation

SUMMARY:
Spontaneous Coronary Artery Dissection (SCAD) is a rare and often misdiagnosed cause of Acute Coronary Syndrome (ACS) affecting predominantly young women without cardiovascular risk factors. There is no definitive evidence on the optimal management of SCAD, but the general approach is conservative.

Unlike established evidence-based rehabilitation programs for ACS and heart failure, no cardiac rehabilitation protocol exists for SCAD.

The aim of the study is to report and detail the cardiac rehabilitation program which was proposed to patients previously included in The Study of the Prevalence Fibromuscular Dysplasia in Patient With Haematoma or Spontaneous Coronary Artery Dissection. (DISCO trial - NCT02799186).

DETAILED DESCRIPTION:
The cardiac rehabilitation program was proposed to the patients presenting with SCAD in each interventional cardiology department, according physician's in charge of the patient decision.

The patient who has undergone a cardiac rehabilitation program following the ACS is included in a retrospective way. The patients are informed about this study by the investigator. After a reflection period, the patient is included.

Details regarding the entrance psychosocial evaluation, the entrance exercise treadmill test, the medications changes during rehabilitation, the training program modalities, the exit exercise treadmill test, and the left ventricular ejection fraction evolution (evaluated by echocardiography) were recorded. The safety for each cardiac rehabilitation program was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient previously recruited in The Study of the Prevalence Fibromuscular Dysplasia in Patient With Haematoma or Spontaneous Coronary Artery Dissection. (DISCO trial - NCT02799186) :

  * Patient over 18 years old
  * Patient with a possible diagnosis of spontaneous coronary dissection defined by:
  * ACS presentation
  * Angiographic signs compatible with a SCAD
  * More or less confirmed by intracoronary imaging (OCT/IVUS) or remote angiographic control (upper to 1 month).
  * Patient with signed informed consent to participate in the DISCO study
  * Subject agreeing to the use of his or her personal data in the form of anonymous coding, including in scientific publications.
* patient who has undergone cardiac rehabilitation following the management of acute coronary syndrome.

Exclusion Criteria:

o Exclusion criteria for the DISCO study :

* Minor patient
* Patients of legal age under protective supervision (guardianship, trusteeship)
* Non affiliation to the French social security system
* Coronary dissection of iatrogenic or traumatic origin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient previsouly recruited in the DISCO Registry with cardiac rehabilitation following the management of acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Safety of the cardiac rehabilitation program | day 0 (inclusion)
  absence/presence of chest pain during cardiac rehabilitation, hospitalization for a cardiac complication during the rehabilitation program

SECONDARY OUTCOMES:
Training program modalities | day 0 (inclusion)
  Medications changes during cardiac rehabilitation program

CONTACTS AND LOCATIONS:
Locations (29):
- France (29):
  - CH Annecy Genevois, Annecy
  - CH Henri Duffaut, Avignon
  - CHU Besançon, Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux, Bordeaux
  - Clinique Convert de Bourg en Bresse, Bourg-en-Bresse
  - CHU de Caen, Caen
  - CH de Cannes, Cannes
  - CH Métropole Savoie, Chambéry
  - CH de Chartres, Chartres
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Simone Veil, Eaubonne
  - Clinique de Fontaine, Fontaine-lès-Dijon
  - CHU de Grenoble Alpes, Grenoble
  - CH Haguenau, Haguenau
  - CHU de la Rochelle, La Rochelle
  - CHU de Limoges, Limoges
  - Hôpital de la Croix Rousse - hospices civils de Lyon, Lyon
  - Hôpital Louis Pradel - Hospices civils de Lyon, Lyon
  - Hôpital privé Jacques Cartier, Massy
  - CHR de Metz-Thionville, Metz
  - GHR Mulhouse et Sud Alsace - Hôpital Emile Muller, Mulhouse
  - C.H.U. de Nîmes, Nîmes
  - Hôpital Bichat-Claude-Bernard, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Universitaire de la Pitié-Salpêtrière, Paris
  - Clinique Saint-Hilaire, Rouen
  - CH de Saint-Brieuc, Saint-Brieuc
  - CHU de Toulouse, Toulouse
  - CHU de Tours-Trousseau, Tours

REFERENCES:
- [Background] Combaret N, Gerbaud E, Derimay F, Souteyrand G, Cassagnes L, Bouajila S, Berrandou T, Range G, Meneveau N, Harbaoui B, Lattuca B, Bouatia-Naji N, Motreff P. National French registry of spontaneous coronary artery dissections: prevalence of fibromuscular dysplasia and genetic analyses. EuroIntervention. 2021 Aug 27;17(6):508-515. doi: 10.4244/EIJ-D-20-01046. PMID 33319763
- [Background] Combaret N, Liabot Q, Deiri M, Lhermusier T, Boiffard E, Filippi E, Roule V, Georges JL, Manzo-Silberman S, Fluttaz A, Marliere S, Souteyrand G, Pereira B, Cassagnes L, Motreff P. Characteristics and Prognosis of Patients With Fibromuscular Dysplasia in a Population of Spontaneous Coronary Artery Dissections (from the French Registry of Spontaneous Coronary Artery Dissections "DISCO"). Am J Cardiol. 2022 Jul 15;175:38-43. doi: 10.1016/j.amjcard.2022.04.007. Epub 2022 May 11. PMID 35562298